CLINICAL TRIAL: NCT06004089
Title: Vaginal Transluminal Endoscopic Sacrocolpopexy: A Minimal Invasive Approach for Pelvic Organ Prolapse
Brief Title: Vaginal Transluminal Endoscopic Sacrocolpopexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Elif Cansu Gundogdu, Specialist doctor, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022/514/222/30
Record Dates: First submitted 2023-08-11; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- V NOTES Sacrocolpopexy arm (Experimental): V-NOTES sacrocolpopexy was performed who met the eligibility criteria and gave written informed consent. Pelvic organ prolapse quantification (POP-Q) scores were evaluated before and 1 month after surgery. Quality of life was evaluated before and 1 month after surgery with the Turkish-validated Pelvic Floor Impact Questionnaire (PFIQ-7) and Pelvic Floor Distress Inventory (PFDI-20).
  Interventions: Procedure: V NOTES Sacrocolpopexy

INTERVENTIONS:
Procedure: V NOTES Sacrocolpopexy — The procedure involved a single-port laparoscopic surgery through the vaginal route, aiming to restore pelvic floor function by suspending the vagina to the anterior longitudinal ligament. The surgical approach differs from conventional methods, as these procedures are conducted through abdominal or vaginal routes without the aid of laparoscopic cameras, However, in our approach, we uniquely combine the widely acknowledged gold standard sacrocolpopexy procedure using vaginal route with laparoscopic camera assistance. No experimental drugs or devices were employed; only the surgical approach was modified.

SUMMARY:
This study aims to evaluate the outcomes of V-NOTES sacrocolpopexy following vaginal hysterectomy, focusing on perioperative and early postoperative results. The impact of V-NOTES sacrocolpopexy on patients' quality of life is investigated using validated assessment tools. Additionally, operative time, complications, pain scores were assessed.

DETAILED DESCRIPTION:
Patients who presented to the obstetrics and gynecology outpatient clinic with complaints related to pelvic organ prolapse, had stage III or IV prolapse according to POP-Q classification, were between 45 and 79 years old, had no contraindications for pneumoperitoneum and Trendelenburg position, and were eligible to perform transvaginal NOTES and gave written informed consent were included in the study. Demographic data, age, medical and surgical history, body mass index (BMI), operation time, preoperative and postoperative haemoglobin levels, perioperative complications and length of hospital stay were collected. Pelvic organ prolapse quantification (POP-Q) scores were evaluated before and 1 month after surgery. Quality of life was evaluated before and 1 month after surgery with the Turkish-validated Pelvic Floor Impact Questionnaire (PFIQ-7) and Pelvic Floor Distress Inventory (PFDI-20).

ELIGIBILITY:
Inclusion Criteria:

* Patients who presented to the obstetrics and gynecology outpatient clinic with complaints related to pelvic organ prolapse, had stage III or IV prolapse according to POP-Q classification, were between 45 and 79 years old, had no contraindications for pneumoperitoneum and Trendelenburg position, and were eligible to perform transvaginal NOTES were included in the study.

Exclusion Criteria:

* Patients with previous pelvic inflammatory disease, deep endometriosis, severe pelvic adhesions, and patients who are at risk of gynecological malignancy and are not suitable for transvaginal surgery were not included in the study.

Ages: 45 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
The impact of V-NOTES sacrocolpopexy on patients' quality of life regarding daily activities and emotional health | 1 month
  The impact of pelvic floor function on daily activities and emotional health of life was evaluated before and 1 month after surgery with the Turkish-validated Pelvic Floor Impact Questionnaire (PFIQ-7). This study aimed to evaluate the outcomes of V-NOTES sacrocolpopexy following vaginal hysterectomy, focusing on perioperative and early postoperative results.
The impact of V-NOTES sacrocolpopexy on patients' quality of life regarding level of discomfort | 1 month
  The level of discomfort associated with symptoms was evaluated before and 1 month after surgery with the Turkish-validated Pelvic Floor Impact Questionnaire (PFIQ-7). This study aimed to evaluate the outcomes of V-NOTES sacrocolpopexy following vaginal hysterectomy, focusing on perioperative and early postoperative results.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Gundogdu, M.D.Dr, Principal Investigator — Kartal Dr. Lutfi Kirdar City Hospital
Locations (1):
- Kartal Dr. Lutfi Kirdar City Hospital, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No